CLINICAL TRIAL: NCT02929745
Title: Elucidating the Fundamental Differences Between HLA-Cw6 Positive and HLA-Cw6 Negative Psoriasis Skin Lesions, With a Comparison to Healthy Skin, at the Single Cell Level of the Infiltrated Immune Cell Types
Brief Title: Single Cell Genomics of Psoriatic Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 15-17769
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Psoriasis
Keywords: immunology, genetics
MeSH Terms: conditions — Psoriasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 HLA-Cw6+ (Experimental): HLA-Cw6+ patients will donate blood and skin samples
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw
- 10 HLA Cw6- (Experimental): HLA-Cw6- patients will donate blood and skin samples
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw
- Healthy Skin (Experimental): Healthy patients will donate blood and skin samples
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw

INTERVENTIONS:
Procedure: Skin biopsy — Four 4-5 mm punch biopsies of the skin
Procedure: Blood draw — Blood will be drawn to test for HLA-cw6 status

SUMMARY:
The purpose of this study is to understand how genetics play a role in psoriasis. Specifically, a genetic allele HLA-Cw6 is known to be associated with psoriasis, and this study aims to find out how it affects genetic and protein expression in patients with psoriasis, compared to healthy people, at a single-cell level using a novel flow cytometry and RNA-sequencing protocol.

ELIGIBILITY:
Inclusion Criteria:

For subjects in the psoriasis group:

1. Ability to provide written consent and comply with the protocol
2. At least 18 years of age
3. Diagnosis of plaque psoriasis for at least 6 months prior to enrollment
4. BSA > 5% and at least one target plaque on trunk or extremities greater than 10cm2

For control subjects:

1. Ability to provide written consent and comply with the protocol
2. At least 18 years of age
3. No previous diagnosis of psoriasis or other inflammatory skin conditions

Exclusion Criteria:

For subjects in the psoriasis group:

1. Subject has non-plaque form of psoriasis.
2. Subject has drug-induced psoriasis.
3. Pregnancy at any point during the study period.
4. Known allergy to lidocaine, other local anesthetics, or any component of local anesthetic agents.
5. Known HIV positive status.
6. Evidence of abnormality of any immune cell population from a drug-induced or genetic cause.
7. Known coagulopathy.

For control subjects:

1. Any physical examination findings by the investigators consistent with psoriasis or other inflammatory skin conditions.
2. Pregnancy at any point during the study period.
3. Known allergy to lidocaine, other local anesthetics, or any component of local anesthetic agents.
4. Known HIV positive status.
5. Evidence of abnormality of any immune cell population from a drug-induced or genetic cause.
6. Known coagulopathy.
7. Use of any immunosuppressant or immunomodulating therapies within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-07-01; Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Determination of immune cell population from skin biopsies | once

SECONDARY OUTCOMES:
Determination of diferentially expressed genes from skin biopsies | once
Determination of HLA -cw6 status from blood samples | once

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Liao, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis Center, San Francisco, California, United States

REFERENCES:
- [Background] Liu J, Chang HW, Huang ZM, Nakamura M, Sekhon S, Ahn R, Munoz-Sandoval P, Bhattarai S, Beck KM, Sanchez IM, Yang E, Pauli M, Arron ST, Fung-Leung WP, Munoz E, Liu X, Bhutani T, North J, Fourie AM, Rosenblum MD, Liao W. Single-cell RNA sequencing of psoriatic skin identifies pathogenic Tc17 cell subsets and reveals distinctions between CD8+ T cells in autoimmunity and cancer. J Allergy Clin Immunol. 2021 Jun;147(6):2370-2380. doi: 10.1016/j.jaci.2020.11.028. Epub 2020 Dec 9. PMID 33309739